CLINICAL TRIAL: NCT06999473
Title: Assess and Treat Visuospatial Neglect in Central Neurological Conditions Via an Innovative Virtual Reality Software
Brief Title: Assessment and Treat Neglect Patients With a VR Application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Wim Saeys, Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241201ACADEM
Record Dates: First submitted 2025-04-27; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Neglect, Hemispatial; Stroke; Virtual Reality Therapy
MeSH Terms: conditions — Perceptual Disorders; Stroke | interventions — Physical Therapy Modalities; Occupational Therapy; Physical Examination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR group (Experimental): The experimental group will receive both conventional OT and PT treatment but 3 days a week, half an hour of conventional treatment will be replaced by treatment with SpatialSense software. The experimental group will receive SpatialSense training 3 times a week for a consecutive 4 weeks (12 sessions in total of 30 minutes).
  Interventions: Device: Virtual reality training; Behavioral: physiotherapy and occupational therapy; Device: Assessment
- Conventional (Active Comparator): The control group will have the assessment on SpatialSense and then receive their regular dose-matched conventional OT and PT sessions without interference. All people with stroke receive conventional occupational (OT) and physical therapy (PT) for 1 hour each. In a total of 4 weeks, 5 times a week.
  Interventions: Behavioral: physiotherapy and occupational therapy; Device: Assessment
- Non-neglect stroke group (Other): Prior to the assessment in SpatialSense, the screen of the head-mounted display will be projected onto a laptop and the eye tracking will be calibrated to the participants' eye positions by the investigator. Then, all participants will perform the assessment part in SpatialSense.
  During assessments with SpatialSense, participants will sit in a wheelchair or on a straight-back chair. The trunk will be restricted to the chair. Finally, the data will be exported from SpatialSense and analyzed by investigators to define different search strategies while performing scanning tasks.
  Interventions: Device: Assessment

INTERVENTIONS:
Device: Virtual reality training — This training is built for the HMD Pico 4 Enterprise, which has six degrees of freedom, a 4k RGB display, a 101-degree field of view, and built-in eye-tracking hardware and software. The virtual environment is a 3-dimensional immersive environment in which the participant will be placed in three different virtual scenes: a picnic table, a kitchen, and a playground. This allows for the placement of stimuli in three different regions: near peripersonal (reaching) space, far peripersonal space, and extrapersonal (far) space. The goal of the game is to search for items that appear in front of the view, as accurately and quickly as possible.
  Arms: VR group
Behavioral: physiotherapy and occupational therapy — The conventional treatment consists of a problem-solving approach mainly based on the neurodevelopmental treatment approach. For VSN, the conventional treatment mainly consists of a mix of prism adaptation, visual scanning, and compensatory strategies based on the individual needs of the patient.
  Arms: Conventional; VR group
Device: Assessment — During assessments with SpatialSense, participants will sit in a wheelchair or on a straight-back chair. The trunk will be restricted to the chair. Finally, the data will be exported from SpatialSense and analyzed by investigators to define different search strategies while performing scanning tasks.

SUMMARY:
The objective of this project is to investigate the effectiveness of neglect training in our self-developed VR application "SpatialSense". The investigators aim to reach the following goals:

i. Compare conventional neglect therapy for neglect training with SpatialSense to evaluate the impacts on neglect recovery to see whether the VR therapy improves the clinical outcomes, such as balance recovery, perception of verticality, quality of life, independence in daily activities, and cognitive impairment, after rehabilitation training.

ii. Analyze and compare the search strategies employed by stroke patients with VSN and those without VSN during the execution of the search task with SpatialSense to summarize typical visual scanning strategies for facilitation, rehabilitation training, and improving the transfer effect in daily activities.

The experimental group will receive both conventional OT and PT treatment, but 3 days a week, half an hour of conventional treatment will be replaced by treatment with SpatialSense software. The control group will receive their regular dose-matched conventional OT and PT sessions without interference. The experimental group will receive SpatialSense training 3 times a week for a consecutive 4 weeks (12 sessions in total of 30 minutes).

DETAILED DESCRIPTION:
Technical information: Our VR application is made with the game engine Unity (version 2020.2.5f1). We built this for the HMD Pico 4 Enterprise, which has six degrees of freedom, a 4K RGB display, a 101-degree field of view, and built-in eye-tracking hardware and software. The virtual environment is a 3-dimensional immersive environment in which the participant will be placed in three different virtual scenes: a picnic table, a kitchen, and a playground. This allows for the placement of stimuli in three different regions: near peripersonal (reaching) space, far peripersonal space, and extrapersonal (far) space. The goal of the game is to search for items that appear in front of the view, as accurately and quickly as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to provide informed consent
3. have had a hemispheric stroke

Exclusion Criteria:

1. Have a severe comorbid psychiatric (E.g. psychotic symptoms) disorder
2. Have a premorbid neurodegenerative disease (E.g. Alzheimer's dementia, vascular dementia)
3. Have severe written language comprehension deficits
4. Have a medical implant, such as a cochlear implant or a pacemaker
5. Have a severe visual impairment that cannot be corrected by wearing glasses while training
6. Have a history of epileptic seizures The following exclusion criteria do not apply to the Non-VSN stroke group.
7. Do not show signs of a spatial asymmetry in performance on a battery of screening tasks
8. Having visual field deficits or lesions in the occipital lobe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in searching performance and visuospatial neglect | Baseline (Day 1) and End of Study (Day 30)
  The Broken Hearts Cancellation Test is a paper-and-pencil assessment used to measure searching performance and spatial neglect. Participants are asked to identify and cancel out complete heart shapes among distractor stimuli (broken hearts) within a fixed time frame. Performance is evaluated based on the number of correct cancellations and errors (false positives and omissions).
  The total score is calculated as:
  Total Correct Hits: Number of correctly cancelled complete hearts (max score: 50) Errors: Number of incorrectly marked broken hearts or missed targets Higher total correct scores indicate better performance. Improvement is defined as an increase in correct hits and/or a reduction in errors.

SECONDARY OUTCOMES:
Change in visuospatial neglect | Baseline (Day 1) and End of Study (Day 30)
  The Schenkenberg Line Bisection Test assesses visuospatial neglect by requiring participants to mark the perceived midpoint of horizontal lines printed on a sheet. The test evaluates the presence and severity of spatial attention deficits, particularly following brain injury or stroke.
  Performance is quantified as the average deviation (in millimeters) from the true midpoint of each line:
  Positive values indicate a rightward deviation Negative values indicate a leftward deviation A score closer to 0 mm indicates better spatial accuracy
Change in functional neglect symptoms | Baseline (Day 1) and End of Study (Day 30)
  The Catherine Bergego Scale (CBS) is a standardized observational tool used to assess the presence and severity of unilateral spatial neglect in activities of daily living. A set of 10 real-life tasks (e.g., grooming, navigating through doorways) will be scored from 0 to 3:
  0 = No neglect
  1. = Mild neglect
  2. = Moderate neglect
  3. = Severe neglect The total score ranges from 0 to 30, with higher scores indicating more severe neglect.
Change in visual search reaction time | Baseline (Day 1) and End of Study (Day 30)
  The Computerized Visual Search Time Test assesses visual attention and processing speed by requiring participants to locate and identify a target stimulus among distractors on a computer screen. The test records the response time (in milliseconds) needed to correctly identify the target.
  Shorter reaction times indicate better visual processing and attention.
Change in spatial and searching performance | Baseline (Day 1) and End of Study (Day 30). Through study completion, an average of 7days
  To assess neglect in our application, we will extract Embedded game parameters from SpatialSense, the maximal rightward angle is compared with the maximal leftward angle on low, medium, and high difficulty levels: the trajectory of the gaze ray (GR), head movement (HR), and eye movement (ER). The maximum angles are added to form the search area middle (SAM) which should be close to 0. A positive SAM indicates the participant searched further to the right than to the left, and a negative SAM means the participant searched further to the left than to the right.
Change in trunk control | Baseline (Day 1) and End of Study (Day 30)
  The Trunk Impairment Scale (TIS) assesses motor impairment of the trunk after neurological injury, especially stroke. It includes three subscales: Static Sitting Balance (0-7); Dynamic Sitting Balance (0-10); Coordination (0-6).
  The total score ranges from 0 to 23, with higher scores indicating better trunk function and postural control.
Change in balance ability | Baseline (Day 1) and End of Study (Day 30)
  The Berg Balance Scale (BBS) is a performance-based measure of balance and fall risk. It consists of 14 functional tasks (e.g., standing up, reaching forward, turning) that are each scored from 0 to 4, based on performance.
  Total score range: 0 to 56. Higher scores indicate better balance. A score below 45 is associated with increased fall risk.

OTHER OUTCOMES:
Change in perceived postural alignment | Baseline (Day 1) and End of Study (Day 30)
  The Subjective Postural Vertical (SPV) test evaluates a person's ability to perceive upright body orientation. During the assessment, the participant is seated on a tilting chair with arms folded across the chest, feet off the ground, and the trunk secured with belts. The head and legs remain free. The examiner tilts the chair at a constant speed of ±1.5°/s. The participant is asked to indicate when they perceive themselves as being in a vertical position.
  Performance is measured in degrees (°) of deviation from true vertical. Lower deviation values indicate better accuracy in vertical perception. Normative values for SPV are approximately 0.12° ± 1.49°.
Change in perceived visual verticality | Baseline (Day 1) and End of Study (Day 30)
  The Subjective Visual Vertical (SVV) test assesses an individual's ability to perceive gravitational vertical using visual cues. In this assessment, participants are seated 1.5 to 2 meters away from a display showing a tilted line. The examiner adjusts the line's angle until the participant indicates that it appears vertically aligned.
  This is commonly administered using the bucket test or a computerized visual display. Performance is measured as the angular deviation (in degrees) from true vertical. Smaller deviations indicate more accurate vertical perception. Normative SVV values typically range between -2.5° and +2.5°.
Change in cognitive function | Baseline (Day 1) and End of Study (Day 30)
  The Mini-Mental State Examination (MMSE) is a widely used 30-point questionnaire that assesses global cognitive function. It evaluates: Orientation, Registration, Attention and calculation, Recall, Language, and Visual construction.
  The total score ranges from 0 to 30, with higher scores indicating better cognitive function. A score below 24 typically suggests cognitive impairment.
Change in quality of life | Baseline (Day 1) and End of Study (Day 30)
  The SS-QOL scale is a patient-centered outcome measure designed to evaluate health-related quality of life in individuals who have experienced a stroke. This self-report instrument consists of 49 items distributed across 12 domains, including energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, cognition, and personality. Each item is rated on a 5-point Likert scale, ranging from 1 (unable to perform the activity, requiring total assistance) to 5 (no difficulty, no assistance required). Higher scores reflect better functional outcomes.
Change in functional independence | Baseline (Day 1) and End of Study (Day 30)
  The FIM is used to assess functional performance in essential daily living skills, including independence in self-care, sphincter control, transfers, mobility, communication, and social cognition. The instrument consists of 18 items, categorized into two subscales: motor and cognitive. Each item is rated on a 7-point ordinal scale, with scores ranging from 1 (total assistance, client expends <25% of the effort) to 7 (complete independence). A higher score indicates a greater level of independence in performing the task related to that item. The total FIM score spans from 18 (complete dependence) to 126 (complete independence).
Change in simulator-induced symptoms | Baseline (Day 1) and End of Study (Day 30)
  The SSQ is a subjective assessment tool used to evaluate the severity of symptoms associated with the use of virtual reality (VR) technology. It comprises 16 items that measure three primary symptom categories: nausea, oculomotor disturbances, and disorientation. The SSQ utilizes a 4-point Likert scale, ranging from 0 (no symptoms) to 3 (severe symptoms), and symptom severity is categorized as negligible (< 5), minimal (5-10), significant (10-15), or concerning (15-20). A total score exceeding 20 is indicative of a "poor " simulator experience.
Change in dynamic balance | Baseline (Day 1) and End of Study (Day 30)
  Mini-BESTest is a quantitative assessment tool for measuring balance and gait functions. It has 14 items, including 4 sections (anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait) with a maximum score of 28. Each item will be rated on a 3-point scale, with 0 indicating severe to 2 indicating normal. Higher scores indicate better balance performance.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Saeys, Study Chair — +32 496804347
Locations (1):
- Rehabilitation Sciences and Physiotherapy, Faculty of Medicine and Health Sciences, University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No